CLINICAL TRIAL: NCT03225638
Title: Performance Evaluation by Magnetic Resonance Imaging (MRI) of Intramuscular Thigh Injections With 3 Configurations of Needle-free Injector (ZENEO®)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CJT-CS-2017-01
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: No Condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Nominal strength thigh injection of 0.65ml of saline solution (0.9%) Low threshold (upper limit) strength thigh injection of 0.65ml of saline solution (0.9%)
  Interventions: Combination Product: Intramuscular ZENEO® injection of nominal strength; Combination Product: Intramuscular ZENEO® injection of low strength (upper limit)
- Group 2 (Other): Nominal strength thigh injection of 0.65ml of saline solution (0.9%) Low threshold (lower limit) strength thigh injection of 0.65ml of saline solution (0.9%)
  Interventions: Combination Product: Intramuscular ZENEO® injection of nominal strength; Combination Product: Intramuscular ZENEO® injection of low strength (lower limit)

INTERVENTIONS:
Combination Product: Intramuscular ZENEO® injection of nominal strength — Sodium Chloride (0.9%)
Combination Product: Intramuscular ZENEO® injection of low strength (upper limit) — Sodium Chloride (0.9%)
  Arms: Group 1
Combination Product: Intramuscular ZENEO® injection of low strength (lower limit) — Sodium Chloride (0.9%)
  Arms: Group 2

SUMMARY:
The aim of this study is to evaluate the intramuscular nominal thigh injection performance and the low threshold strength thigh injection (by evaluating 2 low threshold : upper limit and lower limit). All participants will receive an intramuscular nominal thigh injection, and half of the participants will receive an intramuscular low threshold (upper limit) strength thigh injection, while the other half will receive an intramuscular low threshold (lower limit) strength thigh injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers aged between 18 and 60 years
* Affiliated to or covered by the French social security system
* BMI between ≥ 18 and < 30 kg/m²
* Patients without chronic medical or surgical illness
* Patients with normal clinical examination at the screening visit
* Patients with normal blood pressure at the screening visit: systolic BP < 140 mmHg and diastolic BP < 90 mmHg, determined with the patient seated and resting for at least 5 minutes
* Patient within normal range values for the following laboratory tests (appendix I) unless the investigator considers an abnormality to be clinically irrelevant (to be documented and agreed with the sponsor before inclusion) within 1 month prior to the start of the study.
* Absence of cannabis, opiate, cocaine, amphetamine history
* Written Informed consent

Exclusion Criteria:

* History of drug abuse
* History of hypersensitivity (disease or drug)
* Treatment with platelet inhibiting drugs within one week before inclusion
* Treatment with anticoagulant within four weeks before inclusion
* Subject likely to take any medication during the study
* Contra-indication to MRI: metallic intra-corporeal devices, claustrophobia
* Prior participation to other interventional clinical research within 3 months
* In custody due to administrative or legal decision or under tutelage or being admitted in a sanitary or social institution
* pregnant or breastfeeding woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-12-29 (Estimated)

PRIMARY OUTCOMES:
Depth of the injection | 5 minutes after the injection
  Depth of the injection (mm) by MRI

IPD SHARING:
Plan to Share IPD: Undecided